CLINICAL TRIAL: NCT06057792
Title: Elastography Changes in Cesarean Scar After Negative Pulsed Pressure Treatment
Acronym: ELASTICFLOOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, GONZÁLEZ-MUÑOZ, ANA, PhD Student, MSc, Universidad de Granada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLINICAANAGONZALEZ
Record Dates: First submitted 2023-09-12; First posted 2023-09-28 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Cesarean Scar; Elastography
Keywords: elastography; cesarean; adherences; negative pulsed pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NEGATIVE PULSED PRESSURE INTERVENTION GROUP (Experimental): The number of treatment sessions will consist of a total of 6 sessions, so there will be two sessions over 3 weeks. The evaluations of the participants will be carried out before and after the first session, after the last session of the treatment program received, 15 days and one month after finishing the treatment.
  Interventions: Device: negative pulsed pressure AeroFlow system

INTERVENTIONS:
Device: negative pulsed pressure AeroFlow system — For the application of pulsatile negative pressure, the AeroFlow® equipment will be used, carried out by one of the researchers participating in the project.The application will be carried out addressing the structure of interest (scar), following the protocol established by INDIBA to release adhesions between the different depth planes. The work will consist of an application of pulsed negative pressure using suction cups, which will work automatically at a frequency and intensity tolerable by the patient.
  Treatment protocol in 2 phases Total application time 15min
  1. Static cup: preparation: Prepare the tissue surrounding the scar. 5min
  2. Dynamic Cup: work: Lock the tissue around the scar and the scar itself.10min Suction mode: continuous with continuous sliding of the cup The number of treatment sessions will consist of a total of 6 sessions, so there will be two sessions over 3 weeks.

SUMMARY:
The application of pulsed negative pressure to the scar tissue stimulates the cellular response, producing elastic changes in the tissue, quantifiable by ultrasound, not only in terms of thickness but also in the elastic capacity of the tissues, measured by quantified elastography.

DETAILED DESCRIPTION:
Participants will be recruited at the "Clínica Ana González" physiotherapy clinic. Once recruited, the physiotherapist Ana González Muñoz will carry out the assessment to determine the degree of eligibility of said participants and their inclusion or not in the study. The present study is designed as an open, controlled clinical trial. Two evaluations will be carried out on each participant before and after treatment. Participants who meet the required inclusion/exclusion criteria determined below will be included.

Participants will receive a Negative Pulsed Pressure treatment program with the AeroFlow® equipment. The measuring instruments to be used will be:

- Ultrasound machine.

Description of the ultrasound evaluation

Ultrasound evaluations will be performed. The participant will remain in all measurements. All measurements will be performed with a General Electric S7 R3 The evaluation of tissue quality will be carried out by pixel quantification, using the computer software included in the ultrasound equipment itself.

* Adheremeter Adheremeter is a new device designed to measure postsurgical scar adhesion which is defined as the restriction of scar mobility with respect to the underlying tissue of the point of worst adhesion when stretched in four orthogonal directions. It is an economical and easy-to-use instrument with an ergonomic shape, consisting of 9 concentric rings with radii of 1, 2, 4, 6, 8, 10, 12, 14 and 15 mm, respectively, printed on flexible transparency film for photocopiers. (manufacturer part number PP2500 - 3MTM, St. Paul, MN, USA) to ensure maximum adaptability to different anatomical surfaces.
* Foot posture index (FPI):The foot posture index (FPI) is a reliable instrument for this purpose, assuming a diagnostic tool whose purpose is to quantify the degree of neutral, pronated or supinated position of the foot. The following FPI cut-off points are used, which define the foot type category: a) very supinated from -12 to -4, b) supinated from -3 to 0, c) neutral from 1 to 6, d) pronated from 6 to 10 and e) very pronated from 11 to 12.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 18 and 60 years
* Who have undergone cesarean section surgery and therefore have a scar, lasting more than six months and less than 2 years.
* Patients who present a post-cesarean section scar with a fibrotic appearance and possible surrounding fascial restrictions.

Exclusion Criteria:

* Patients who present any neurological, inflammatory or orthopedic injury that prevents or alters balance, listening, vision or the cognitive abilities necessary to be able to answer appropriate questions or take questionnaires.
* Patients who present keloids in the scar.
* Patients who have contraindications to be treated with a 448kHz radiofrequency device such as:

to. pregnant women b. Subjects with any type of electronic implants. c. Subjects presenting with thrombophlebitis

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2024-02-11 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
elastography measurement | Time0 (T0) FIRST DAY BEFORE FIRST TREATMENT, TIME 1 (T1) FIRST DAY AFTER FIRST TREATMENT, TIME 2 (T2) AFTER 6 DAY OF TREATMENT (THE THIRD WEEK) , TIME 3(T3) 15 DAYS AFTER THE SIXTH TREATMENT, TIME 4 (T4) ONE MONTH AFTER THE SIXTH TREATMENT.
  The elastography is obtained when the anatomic image on grayscale ultrasound overlaps parametric color image that expresses the rate of deformity of the tissues, soft tissues tend to develop greater deformity and tissue deformity have lower rigidity.

SECONDARY OUTCOMES:
adheremeter measurement | Time0 (T0) FIRST DAY BEFORE FIRST TREATMENT, TIME 1 (T1) FIRST DAY AFTER FIRST TREATMENT, TIME 2 (T2) AFTER 6 DAY OF TREATMENT (THE THIRD WEEK) , TIME 3(T3) 15 DAYS AFTER THE SIXTH TREATMENT, TIME 4 (T4) ONE MONTH AFTER THE SIXTH TREATMENT.
  Adheremeter is a new device designed to measure postsurgical scar adhesion which is defined as the restriction of scar mobility with respect to the underlying tissue of the point of worst adhesion when stretched in four orthogonal directions. It is an economical and easy-to-use instrument with an ergonomic shape, consisting of 9 concentric rings with radii of 1, 2, 4, 6, 8, 10, 12, 14 and 15 mm, respectively, printed on flexible transparency film for photocopiers. (manufacturer part number PP2500 - 3MTM, St. Paul, MN, USA) to ensure maximum adaptability to different anatomical surfaces.
Foot posture index | Time0 (T0) FIRST DAY BEFORE FIRST TREATMENT, TIME 1 (T1) FIRST DAY AFTER FIRST TREATMENT, TIME 2 (T2) AFTER 6 DAY OF TREATMENT (THE THIRD WEEK) , TIME 3(T3) 15 DAYS AFTER THE SIXTH TREATMENT, TIME 4 (T4) ONE MONTH AFTER THE SIXTH TREATMENT.
  The foot posture index (FPI) is a reliable instrument for this purpose, assuming a diagnostic tool whose purpose is to quantify the degree of neutral, pronated or supinated position of the foot. The following FPI cut-off points are used, which define the foot type category: a) very supinated from -12 to -4, b) supinated from -3 to 0, c) neutral from 1 to 6, d) pronated from 6 to 10 and e) very pronated from 11 to 12.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Ana González, Málaga
  - Clínica Ana González, Málaga

IPD SHARING:
Plan to Share IPD: Undecided